CLINICAL TRIAL: NCT02295423
Title: A Long-Term Follow-Up Study to Assess Implementation of Ultrasound-Guided Regional Anesthesia Skills Training by Practicing Anesthesiologists
Brief Title: Follow-Up Study to Assess Implementation of Ultrasound-Guided Regional Anesthesia Skills
Status: Completed | Type: Observational
Sponsor: VA Palo Alto Health Care System (U.S. Federal Agency)
Responsible Party: Principal Investigator, Edward R. Mariano, Chief, Anesthesiology and Perioperative Care Service and Associate Chief of Staff for Inpatient Surgical Services VA Palo Alto Health Care System, VA Palo Alto Health Care System
Other Study IDs: 29837
Record Dates: First submitted 2014-10-27; First posted 2014-11-20 (Estimated); Last update posted 2015-12-10 (Estimated); Status verified 2015-12

CONDITIONS: Implementation of Anesthesiologists' Practice Change

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
The investigators hope to survey anesthesiologists who have participated in a non-CME regional anesthesia workshop at VAPAHCS over the past 4 years on the number and types of nerve block procedures that they performed, nerve localization method (e.g., ultrasound, electrical stimulation, or both), and whether the nerve blocks performed were single-injection or catheter-based.

DETAILED DESCRIPTION:
The investigators expect to recruit approximately 100 participants through the use of an IRB-approved survey and cover letter which will be distributed to anesthesiologists who have participated in a non-CME regional anesthesia workshop at VAPAHCS over the past 4 years. Prospective subjects will provide consent to participate by completing the requested survey. Subjects will not receive monetary remuneration for their participation. Selection for inclusion will not be based on gender, race, or socioeconomic status. There will be no recruitment of participants from vulnerable populations. Participants will receive a link to an online survey and if they prefer an alternate method, the investigators will send the participant the survey in Word document format or survey by telephone. The survey will ask for the number and types of nerve block procedures that the participant performed, nerve localization method (e.g., ultrasound, electrical stimulation, or both), and whether the nerve blocks performed were single-injection or catheter-based.

ELIGIBILITY:
Inclusion Criteria: Anesthesiologists in practice who have participated in a regional anesthesia workshop at VAPAHCS; and willingness to complete a survey.

Exclusion Criteria: Anesthesiologists who have visual, hearing, or other communication impairment that would interfere with survey completion.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: We intend to enroll approximately 100 subjects (one site only) based on the estimated number of practicing anesthesiologists who have participated in a regional anesthesia workshop at VAPAHCS within the last 4 years. Subjects who are practicing anesthesiologists out of residency and will likely be 40-70 years of age. We expect to recruit subjects of both genders and all ethnic backgrounds.
Sampling Method: Probability Sample
Enrollment: 99 (Actual)
Dates: Start 2014-11; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Implementation of Ultrasound-Guided Regional Anesthesia skills | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- VA Palo Alto Health Care System, Palo Alto, California, United States

REFERENCES:
- [Background] 1. Sites BD, Spence BC, Gallagher JD, Wiley CW, Bertrand ML, Blike GT. Characterizing novice behavior associated with learning ultrasound-guided peripheral regional anesthesia. Reg Anesth Pain Med2007;32:107-15. 2. Ajmal M, Power S, Smith T, Shorten GD. Ergonomic task analysis of ultrasound-guided femoral nerve block: a pilot study. J Clin Anesth 2011;23:35-41. 3. Ilfeld BM, Enneking FK. Continuous peripheral nerve blocks at home: a review. Anesth Analg 2005;100:1822-33. 4. Ilfeld BM. Continuous peripheral nerve blocks: a review of the published evidence. Anesth Analg 2011;113:904-25. 5. Ilfeld BM, Gearen PF, Enneking FK, Berry LF, Spadoni EH, George SZ, Vandenborne K. Total knee arthroplasty as an overnight-stay procedure using continuous femoral nerve blocks at home: a prospective feasibility study. Anesth Analg 2006;102:87-90. 6. Ilfeld BM, Mariano ER, Williams BA, Woodard JN, Macario A. Hospitalization costs of total knee arthroplasty with a continuous femoral nerve block provided only in the hospital versus on an ambulatory basis: a retrospective, case-control, cost-minimization analysis. Reg Anesth Pain Med 2007;32:46-54. 7. Ramlogan R, Manickam B, Chan VW, Liang L, Adhikary SD, Liguori GA, Hargett MJ, Brull R. Challenges and training tools associated with the practice of ultrasound-guided regional anesthesia: a survey of the American society of regional anesthesia and pain medicine. Reg Anesth Pain Med 2010;35:224-6. 8. Hadzic A, Vloka JD, Kuroda MM, Koorn R, Birnbach DJ. The practice of peripheral nerve blocks in the United States: a national survey [p2e comments]. Reg Anesth Pain Med 1998;23:241-6. 9. Kopacz DJ, Neal JM. Regional anesthesia and pain medicine: residency training--the year 2000. Reg Anesth Pain Med 2002;27:9-14. 10. Kopacz DJ, Neal JM, Pollock JE. The regional anesthesia